CLINICAL TRIAL: NCT03088475
Title: A Randomised Controlled Trial on a Nurse-led Smartphone-based Self-management Programme for Type 2 Diabetes Patients With Poor Glycaemic Control
Brief Title: A Nurse-led Smartphone-based Self-management Programme for Type 2 Diabetes Patients With Poor Blood Glucose Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University of Singapore (Other)
Collaborators: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Wang Wenru, Principal Investigator, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AcRFTier1FRCT1-2016APR-02
Record Dates: First submitted 2017-03-13; First posted 2017-03-23 (Actual); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Type2 Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): A six-month nurse-led smartphone-based self-management programme (i.e. NSSMP) will be provided to the participants in the experimental group.
  Interventions: Behavioral: nurse-led smartphone-based self-management programme
- Control Group (Active Comparator): the patients in the control group will receive the exiting nurse-led diabetes service (i.e. NDS) provided by the hospital
  Interventions: Behavioral: exiting nurse-led diabetes service

INTERVENTIONS:
Behavioral: nurse-led smartphone-based self-management programme — The participants in the experimental group will undergo nurse-led smartphone-based self-management programme (NSSMP), a 6-month programme comprising an individual education session, and a newly developed smartphone App as a self-help education resource
  Arms: Experimental Group
Behavioral: exiting nurse-led diabetes service — the patients in the control group will receive the exiting nurse-led diabetes service (i.e. NDS) provided by the hospital
  Arms: Control Group

SUMMARY:
Aim. To develop and compare a nurse-led smartphone-based self-management programme with an existing nurse-led diabetes service on health-related outcomes of type 2 diabetes patients with poor glycaemic control in Singapore.

Background. Over the past decades, Asia has emerged as the 'diabetes epicentre' in the world due to rapid economic development, urbanisation, and nutrition transition. There is an urgent need to develop more effective care management strategies in response to this rising diabetes epidemic.

Design. A randomised controlled trial with pre- and repeated post-tests control group design.

Methodology. A total of 128 type 2 diabetes patients with poor glycaemic control will be recruited from the diabetes clinic of a public acute hospital in Singapore through convenience sampling. Study participants will be randomly allocated either to the experimental group or the control group. Outcome measures will include the 10-item General Self-Efficacy Scale, 11-item Revised Summary of Diabetes Self-care Activities, and 19-item Diabetes-Dependent Quality of Life. Data will be collected at three time points: baseline, 3 months, and 6 months from the baseline.

Discussion. It is expected that this programme will be an alternative offered to diabetes patients to master their self-care management skills, in addition to the existing diabetes service provided in diabetes clinics in Singapore hospitals. Furthermore, the self-supporting and less resource-intensive nature of this programme, through the use of a smartphone application as the mode of intervention delivery, will greatly reduce nurses' direct contact time with patients and allow more time to be allocated to those who require more attention.

DETAILED DESCRIPTION:
Specific Aims

The aims of this study are:

1. to develop a nurse-led smartphone-based self-management programme (NSSMP) for patients with type 2 diabetes;
2. to compare the NSSMP with an existing nurse-led diabetes service (NDS) on self-efficacy, diabetes self-care activities, health-related quality of life (HRQoL), glycaemic control, acute diabetes complications (e.g. hypoglycaemia, Diabetic Ketoacidosis [DKA] and Hyperosmolar Hyperglycemic Syndrome [HHS]), and health-service use among type 2 diabetes patients with poor glycemic control in Singapore.

Study Hypotheses

Study participants will be randomized into an existing NDS group (i.e. control group) and a newly developed NSSMP group (i.e. experimental group). It is hypothesized that participants in the NSSMP group as compared with participants in the NDS group will have significantly:

1. Higher level of self-efficacy;
2. Increased level of diabetes self-care activities;
3. More positive perceived health-related quality of life;
4. Reduced glycosylated haemoglobin (HbA1c) and acute diabetes complications (e.g. hypoglycaemia, Diabetic Ketoacidosis [DKA] and Hyperosmolar Hyperglycemic Syndrome [HHS] ); and
5. Reduced usage of health services (e.g. diabetes-related hospital readmission, emergency room attendance, and unplanned medical consultation).

Approach Adopted in This Study Development of NSSMP: A nurse-led smartphone-based self-management programme, or NSSMP for short, will be developed by the study team. The model of self-efficacy will be used to guide the development of the NSSMP to ensure it would be theoretically sound and empirically tested. The NSSMP is a 6-month programme comprising an individual education session, and a newly developed smartphone App as a self-help education resource. The NSSMP involves the use of a smartphone, internet, and communication technologies to assist patients to manage their disease at homes or wherever they are. Patient's health data will be monitored by their smartphones. All the data will be synchronized to a web-connected portal on a remote server. The nurse would be able to access the participant's data (e.g. blood glucose, exercise, blood pressure, body weight, diet) through the web-connected portal so that the individualized care and consultation could be rendered through the tele or video conference.

Study design, setting and participants: A randomized controlled trial with a pre- and repeated post-test control group design is adopted. A convenience sample of 128 type 2 DM patients with poor glycemic control will be recruited from the Diabetes Clinic of National University Hospital (NUH). Study participants will be randomly assigned either to a 6-month NSSMP group (i.e experimental group) or the NDS group (i.e. control group). The existing NDS for DM patients in the NUH consists of face-to-face patient education sessions plus telephone follow-ups. The patients are required to return back to the Diabetes Clinic to attend the educations sessions based on the scheduled appointment. They are instructed to measure blood glucose at home and modes of contact (voicemail, fax and email address) are given for reporting the glucose readings weekly. If the patient does not report, the nurse will have to make calls or send SMS message to the patient to follow up their blood glucose results. The nurses would then provide telephone counselling services to the patients where needed based on the blood glucose results, and sometime would request patients coming back to the Diabetes Clinic to see the doctors and the diabetes advanced practice nurses.

Outcome measures: Study outcome measures include the 10-item General Self-Efficacy Scale, 11-item Revised Summary of Diabetes Self-care Activities, and 19-item Diabetes-Dependent Quality of Life which will be used to measure self-efficacy, level of diabetes self-care activities, and health-related quality of life of the participants respectively. The participant's socio-demographic and clinical data (e.g. HbA1c, acute diabetes complications, and lipid level) will be also collected. Data will be collected at 3 time points: baseline (i.e. pre-test), 3 months from baseline (post-test 1), and 6 months from the baseline (post-test 2). The health service use (e.g. diabetes-related hospital readmission, emergency room attendance, and unplanned medical consultation) will be also assessed at the 6th month of the end of the programme.

Data analysis: The IBM SPSS 23.0 will be used for data entry and analysis. Intention-to-treat will be adopted in data analysis. Repeated measures analysis of covariance will be used to examine the differences between, within, and the interaction (group x time) effects on each continuous outcome. Confounding variables (e.g. age), will be controlled as covariate in the analysis. The Chi-squared test or Fisher's exact test will be used to test the difference of the incidence of acute diabetes complications and the numbers of health service use between the two groups. All statistical tests will be two-tailed, and a p < 0.05 is used to indicate statistical significance.

Study Significance If the NSSMP is demonstrated to be effective in this study, a smartphone App developed in this project can be provided to all DM patients and their family members/caregivers as a self-help education resource at home. It will provide and equip knowledge to the patient and their family members/caregivers to enhance their knowledge and skills in management of diabetes so as to achieve the expected patient outcomes in improving self-efficacy, diabetes self-care activities, HRQoL, and clinical outcomes. It is expected that this programme will be an option that can be offered to diabetes patients to master their self-care management skills in addition to the existing diabetes service provided in diabetes clinics in Singapore hospitals where patients with poorly controlled condition are being monitored. In addition, the independent nature of this programme with application of technology will greatly reduce nurses' contact time with patients which accord them more time for those who require more time, for example, those afflicted with diabetes-related complications. This will result in a more efficient use of healthcare resources in the long run. Eventually, this programme will be available for all diabetes patients living in the community.

Feasibility of the Study The research team comprises experienced researchers from different disciplines. The PI has extensive research experience in the area of chronic diseases management and mHealth intervention. Two Co-Is are practised clinicians in diabetes care, they will facilitate the access to potential study participants and oversee the implementation of the project. One Co-I has the expertise in biomedical engineering, mobile App development, and information management. He and his team will be in charge of developing the system. In addition, the preliminary integrative literature review and qualitative patient interviews were performed to inform the development of the content for the mobile app. Through harnessing the technology, the smartphone App based platform can be established to reduce the contact time with patients for the healthcare providers.

ELIGIBILITY:
Inclusion Criteria:

* have confirmed medical diagnosis of type 2 DM;
* are 21 years old and above;
* have blood test result of HbA1c > 8% in the most recent test indicating poor glycemic control;
* possess and able to use smart mobile phone (e.g. Samsung Galaxy, iPhone) in their daily lives; and
* are able to speak and read English or Chinese.

Exclusion Criteria:

* have suffered severe complications such as severe stroke, visual impairment, renal failure that interfere with self-care activities;
* have known history of major psychiatric illness;
* have reading and hearing difficulties.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Self-efficacy: change is being assessed | Change from baseline self-efficacy at 6 months
  Self-efficacy will be assessed using the General Self-efficacy Scale (GSS), a 10-item questionnaire of the unidimensional measure of one's competence to deal with the challenging events encountered in various life situations

SECONDARY OUTCOMES:
Diabetes self-care activities: change is being assessed | Change from baseline diabetes self-care acitivities at 6 months
  Diabetes self-care activities will be measured using the 11-item Revised Summary of Diabetes Self-care Activities (RSDSCA)
Health-related Quality of Life: change is being assessed | Change from baseline health-related quality of life at 6 months
  Health-related Quality of Life will be measured using the 19-item Diabetes-Dependent Quality of Life (DDQoL)
Acute Diabetes Complications: change is being assessed | Change from baseline acute diabetes complications at 6 months
  the number of frequency of acute diabetes complications including hypoglycaemia, DKA and HHS will be collected
HbA1c: change is being assessed | Change from baseline HbA1c at 6 months
  HbA1c will be obtained from patient's medical record
Smoking status: change is being assessed | Change from baseline smoking status at 6 months
  Smoking status will reported by the participant.
Alcohol consumption: change is being assessed | Change from baseline alcohol consumption at 6 months
  Alcohol consumption will be reported by the participant
Diabetes-related hospital admission | at the 6-month of the study period
  number of diabetes-related hospital admission will be recorded
Visits to the emergency | at the 6-month of the study period
  number of diabetes-related emergency department visit will be recorded
Unplanned medical consultation | at the 6-month of the study period
  number of unplanned medical consultation due to diabetes problems will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Wenru P Wang, PhD, Principal Investigator — National University of Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jiang Y, Ramachandran HJ, Teo JYC, Leong FL, Lim ST, Nguyen HD, Wang W. Effectiveness of a nurse-led smartphone-based self-management programme for people with poorly controlled type 2 diabetes: A randomized controlled trial. J Adv Nurs. 2022 Apr;78(4):1154-1165. doi: 10.1111/jan.15178. Epub 2022 Feb 15. PMID 35170786
- [Derived] Wang W, Seah B, Jiang Y, Lopez V, Tan C, Lim ST, Ren H, Khoo YH. A randomized controlled trial on a nurse-led smartphone-based self-management programme for people with poorly controlled type 2 diabetes: A study protocol. J Adv Nurs. 2018 Jan;74(1):190-200. doi: 10.1111/jan.13394. Epub 2017 Aug 17. PMID 28727183